CLINICAL TRIAL: NCT03227484
Title: A Double-blind Randomized Study to Determine the Effect of Empagliflozin Versus Placebo on Brain Insulin Sensitivity in Patients With Prediabetes
Brief Title: Effect of Empagliflozin Versus Placebo on Brain Insulin Sensitivity in Patients With Prediabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Empabrain01
Record Dates: First submitted 2017-06-07; First posted 2017-07-24 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2019-07

CONDITIONS: PreDiabetes; Body Weight
MeSH Terms: conditions — Prediabetic State; Body Weight | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin (Active Comparator): 25mg Empagliflozin once daily over 8 weeks
  Interventions: Drug: Empagliflozin 25mg
- Placebo (Placebo Comparator): Matching placebo tablet once daily over 8 weeks
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Empagliflozin 25mg — Once daily over 8 weeks
  Arms: Empagliflozin
Drug: Placebo Oral Tablet — Once daily over 8 weeks
  Arms: Placebo

SUMMARY:
Recently, various sodium glucose cotransporter 2 (SGLT2) inhibitors have been approved for the treatment of type 2 diabetes mellitus. Empagliflozin is a preparation of this class of substances. SGLT2 inhibitors also lead to a reduction in body weight in addition to their blood glucose lowering effect. The basis for this is probably the calorie loss by the increased glucose excretion over the urine. However, this weight-reducing effect is lost after a few weeks of treatment and the body weight subsequently stabilizes at a lower level than before. However, patients continue to lose energy via the urine. Hence, the weight stabilization could be due to an increased energy intake as a possible consequence of a changed brain setpoint for the body weight. As the main weight loss is achieved during the first 6-8 weeks of treatment, the investigators assume that the underlying central nervous mechanisms will be present after this time.

Furthermore, clinical-experimental observations show that treatment with empagliflozin promotes endogenous glucose production in the liver. This presumably compensatory mechanism also occurs after only a few weeks of treatment. The common mechanism, which could be based both on energy intake and on the endogenous glucose production effect, is still unclear. The investigators suspect that regulatory circuits in the brain contribute to these observed effects.

In fact, several studies in animals as well as initial clinical studies in humans show that the brain is involved in eating behavior and peripheral metabolism. In particular, effects of the hormone insulin modulate the dietary intake via the brain, thereby affecting human body weight.

Many of the experiments on the insulin sensitivity of the human brain used a specific approach to the selective delivery of insulin into the brain: the application of insulin as a nasal spray. Although this application route has no therapeutic value, this technique allows the administration of insulin to the central nervous system with little effect on the circulating insulin levels. By combining nasal insulin administration with functional MRI, regional insulin sensitivity of the brain can be quantified. The investigators recently found that the insulin action of the brain (stimulated by nasal insulin) regulates both endogenous glucose production and peripheral glucose uptake during hyperinsulinemic euglycemic glucose clamps. The signals from the brain seem to reach the periphery via the autonomic nervous system in order to modulate metabolic processes. A central brain area in this regard is the hypothalamus. This brain region receives afferents over various systems such as the autonomic nervous system and various endocrine systems (including insulin). The investigators recently characterized the hypothalamus as an insulin-sensitive brain area in humans. The hypothalamus is the key area for homeostatic control throughout the body.

Since the dietary intake and the endogenous glucose production are modulated by a hypothalamic insulin effect in humans, we suspect that the observed effects of SGLT2 inhibitors on both processes could be due to altered insulin activity in the brain. Since the SGLT2 inhibition by empagliflozin modulates the autonomic nervous system in the kidneys, signals from the kidney may be transmitted to the brain via the autonomic nervous system, thereby changing specific setpoints, including e.g. insulin sensitivity of the brain.

In order to test this hypothesis, a precise phenotyping of prediabetic volunteers with regard to regional brain insulin sensitivity as well as the brain effect on metabolism before and after 8 weeks of treatment with empagliflozin compared to placebo is planned.

ELIGIBILITY:
Inclusion Criteria:

* Fasting blood glucose between 100 and 125 mg/dl and/or 2-hour post load glucose between 140 and 199 mg/dl during a 75 g oral glucose tolerance test.
* Body mass index (BMI) between 25 and 40 kg/m².
* Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures.
* Ability to adhere to the study visit schedule and other protocol requirements.
* Females of childbearing potential (FCBP1) must agree
* to utilize two reliable forms of contraception simultaneously or practice complete abstinence from heterosexual contact for at least 28 days before starting study drug, while participating in the study (including dose interruptions), and for at least 28 days after study treatment discontinuation and must agree to pregnancy testing during this timeframe
* to abstain from breastfeeding during study participation and 28 days after study drug discontinuation.
* Males must agree
* to use a latex condom during any sexual contact with FCBP while participating in the study and for 28 days following discontinuation from this study, even if he has undergone a successful vasectomy
* to refrain from donating semen or sperm while participating in this study and for 28 days after discontinuation from this study treatment.
* All subjects must agree to refrain from donating blood while on study drug and for 28 days after discontinuation from this study treatment.
* All subjects must agree not to share medication.

Exclusion Criteria:

* Women during pregnancy and lactation.
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal products. This includes empagliflozin, placebo and human insulin.
* Participation in other clinical trials or observation period of competing trials up to 30 days prior to this study.
* Diabetes mellitus
* Known malformation of the central nervous system
* Persons working nightshift
* Treatment with glucose lowering drugs, drugs with central nervous actions or systemic steroid therapy
* Any relevant (according to investigator's judgment) cardiovascular disease, e.g. myocardial infarction, acute coronary syndrome, unstable angina pectoris, Percutaneous transluminal coronary angioplasty (PTCA), heart failure (NYHA II-IV), stroke or transient ischemic attack (TIA), within 12 months prior to screening.
* Indication of liver disease, as per medical history or defined by serum levels of either Alanine Aminotransferase (ALT [SGPT]), Aspartate Aminotransferase (AST [SGOT]), or alkaline phosphatase above 3 x upper limit of normal (ULN) as determined during screening.
* Alcohol abuse, defined as more than 20 gr/day
* Impaired renal function, defined as estimated Glomerular Filtration Rate (eGFR) ≤ 60 ml/min (MDRD formula) as determined during screening.
* Known structural and functional urogenital abnormalities, that predispose for urogenital infections.
* Subjects with a haemoglobin (Hb) ≤ 11.5 g/dl (for males) and Hb ≤ 10.5 g/dl (for females) at screening.
* Bariatric surgery within the past two years and other gastrointestinal surgeries that induce chronic malabsorption within the last 5 years.
* Medical history of cancer (except for basal cell carcinoma) and/or treatment for cancer within the last 5 years.
* Treatment with anti-obesity drugs 3 months prior to informed consent or any other treatment at the time of screening (i.e. surgery, aggressive diet regimen, etc.) leading to unstable body weight.
* Known autoimmune disease (except autoimmune disease of the thyroid gland) or chronic inflammatory condition.
* Claustrophobia
* Any other clinically significant major organ system disease at screening such as relevant gastrointestinal, neurologic, psychiatric, endocrine (i.e. pancreatic), hematologic, malignant, infection or other major systemic diseases making implementation of the protocol or interpretation of the study results difficult.
* Presence of any contraindication for the conduct of an MRI investigation, such as cardiac pacemakers, ferromagnetic haemostatic clips in the central nervous system, metallic splinters in the eye, ferromagnetic or electronically operated active devices like automatic cardioverter defibrillators, cochlear implants, insulin pumps and nerve stimulators, prosthetic heart valves etc.
* Refusal to get informed of unexpected detected pathological MRI findings

Any other clinical condition that would jeopardize subjects' safety while participating in this clinical trial.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
effect of treatment with 25 mg empagliflozin daily versus placebo on regional brain insulin sensitivity | baseline and after 8 weeks of treatment
  assessed by functional magnetic resonance imaging (fMRI) combined with nasal insulin administration as change from baseline to 8 weeks

SECONDARY OUTCOMES:
effects of treatment with empagliflozin versus placebo on glucose tolerance in prediabetes | baseline and after 8 weeks of treatment
  assessed by 75g oral glucose tolerance test (oGTT) as change from baseline to 8 weeks
effects of treatment with empagliflozin versus placebo on body fat composition | baseline and after 8 weeks of treatment
  assessed by whole body MRI and liver MR-spectroscopy and bioimpedance analysis as change from baseline to 8 weeks
effect of treatment with empagliflozin versus placebo on brain-insulin derived modulation of peripheral metabolism | baseline and after 8 weeks of treatment
  assessed by hyperinsulinemic euglycemic clamp combined with nasal insulin administration as change from baseline to 8 weeks
effect of treatment with empagliflozin versus placebo on autonomous nervous system activity | baseline and after 8 weeks of treatment
  assessed by analysis of heart rate variability as change from baseline to 8 weeks
effect of treatment with empagliflozin versus placebo on the brain responsiveness to food cues and nutrient-specific food preference | baseline and after 8 weeks of treatment
  assessed by fMRI combined with nasal insulin administration as change from baseline to 8 weeks
effect of treatment with empagliflozin versus placebo on the correlation between insulin secretion capacity and regional brain insulin sensitivity | baseline and after 8 weeks of treatment
  assessed by fMRI combined with nasal insulin administration and 75g oGTT as change from baseline to 8 weeks
effect of treatment with empagliflozin versus placebo on energy expenditure | baseline and after 8 weeks of treatment
  assessed by indirect calorimetry as change from baseline to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martin Heni, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University of Tuebingen, Department of Internal Medicine IV, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hummel J, Machann J, Dannecker C, Kullmann S, Birkenfeld AL, Haring HU, Peter A, Fritsche A, Wagner R, Heni M. Eight weeks of empagliflozin does not affect pancreatic fat content and insulin secretion in people with prediabetes. Diabetes Obes Metab. 2022 Aug;24(8):1661-1666. doi: 10.1111/dom.14733. Epub 2022 Jun 6. No abstract available. PMID 35475570
- [Derived] Kullmann S, Hummel J, Wagner R, Dannecker C, Vosseler A, Fritsche L, Veit R, Kantartzis K, Machann J, Birkenfeld AL, Stefan N, Haring HU, Peter A, Preissl H, Fritsche A, Heni M. Empagliflozin Improves Insulin Sensitivity of the Hypothalamus in Humans With Prediabetes: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Trial. Diabetes Care. 2022 Feb 1;45(2):398-406. doi: 10.2337/dc21-1136. PMID 34716213